CLINICAL TRIAL: NCT00654355
Title: Measuring Adherence to Topical Therapy in Children With Atopic Dermatitis and the Impact of a Return Visit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002300; contract #32417 (Other: WakeForest)
Record Dates: First submitted 2008-04-02; First posted 2008-04-08 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Drug (Experimental): tacrolimus ointment
  Interventions: Drug: tacrolimus ointment

INTERVENTIONS:
Drug: tacrolimus ointment — tacrolimus ointment to be applied twice daily to affected areas during duration of study
  Other Names: Protopic Ointment

SUMMARY:
The purpose of this research study is to better understand how the study drug works when people use it to treat atopic dermatitis.

DETAILED DESCRIPTION:
To evaluate adherence to topical therapy using adherence data collected by the MEMS cap (Medication Electronic Monitoring System) in pediatric patients with atopic dermatitis (AD) and the impact of a return visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age 2-15.
2. Stable or worsening atopic dermatitis affecting 5% or greater body surface area. Face and genital areas can be included in the body surface area determination and treatment area.
3. The ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study.
4. The ability to understand and sign a written informed consent/assent form, which must be obtained prior to treatment.

Exclusion Criteria:

1. Known allergy to tacrolimus or to any component of the formulations.
2. The use of systemic therapy for atopic dermatitis within the past 4 weeks.
3. Use of prescription topical therapy for atopic dermatitis (e.g., corticosteroids or retinoids) within the past 2 weeks.
4. Use of any investigational therapy within the past 4 weeks.
5. Pregnant females, females who are breast feeding, or females of childbearing potential who are not practicing an acceptable method of birth control (abstinence, birth control pill/patch, barrier with spermicidal jelly, IUD, etc.), as determined by the investigator. Acceptable contraception must be used during the entire study. A pregnancy test will be performed on females of childbearing potential at baseline and at week 4.
6. Any other condition which, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Feldman, MD, PHD, Principal Investigator — WFUHS
Locations (1):
- Dept of Dermatology, WFUHS, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Dermatology Studies Center and IRB approved advertising.
Groups:
- Control Group: Group only had visits at Baseline and Week 4.
- Extra Visit Group: After Baseline, this group had an extra visit at week 1.
Period: Overall Study
Arm/Group | Control Group | Extra Visit Group
Started | 15 | 15
Completed | 13 | 13
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Extra Visit Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: adherence to topical therapy in children via MEMS cap in a "real-life" clinic population measured as the % of required applications completed
Time Frame: Week 4
Measure: Median (95% Confidence Interval); unit: percentage of required applicaitons
Arm/Group | Control Group | Extra Visit Group
Number analyzed (Participants) | 15 | 15
percentage of required applicaitons | 56 [15 to 79] | 72 [39 to 114]

2. Secondary Outcome: The % Change From Baseline to Week 4 (or End of Treatment) in the IGA.
Description: Investigator Global Assessment: Investigator's Global Assessment of severity integrates all lesions for overall score. This measure is commonly used as a quick and simple way to quantify disease severity both for clinical studies and in a non-study clinic setting. Score ranges from '0' = clear or "No inflammatory signs of AD" to '4' = Very Severe Disease with "severe erythema and severe papulation/infiltration with oozing/crusting."
Time Frame: Week 4
Measure: Median (95% Confidence Interval); unit: % change in IGA
Arm/Group | Control Group | Extra Visit Group
Number analyzed (Participants) | 15 | 15
% change in IGA | -33 [-44 to -18] | -33 [-54 to -30]

3. Secondary Outcome: EASI
Description: Eczema Area and Severity Index (EASI): Disease severity will be assessed by a physician with the Eczema Area and Severity Index (EASI). This measure is commonly used and well validated instrument of eczema severity. It is weighted for area in each of the four body regions (which differs for adults and children under 7) and scores erythema, excoriation, induration/papulation, and lichenification. The total scores range from 0-72. Higher scores represent more severe eczema.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Extra Visit Group
Number analyzed (Participants) | 15 | 15
units on a scale | 2.1 (5.7) | 1 (2.6)

ADVERSE EVENTS:
Arm/Group | Control Group | Extra Visit Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=15) | Extra Visit Group (N=15)
Upper respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No